CLINICAL TRIAL: NCT06904287
Title: Evaluating the Effectiveness of Magnesium in Addition to Prochlorperazine for the Treatment of Migraines in the Emergency Department
Brief Title: Effectiveness of Magnesium in Addition to Prochlorperazine for the Treatment of Migraines
Acronym: MAGraine2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00127959
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Migraine; Magnesium
MeSH Terms: conditions — Migraine Disorders | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Drug (Experimental): Prochlorperazine 10 mg followed by Magnesium 2 g
  Interventions: Drug: Magnesium
- Control Arm (Active Comparator): Prochlorperazine 10 mg followed by placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium — Prochlorperazine 10 mg administered as an intravenous push over 2 minutes followed by magnesium 2 g administered as an intravenous bolus over a period of 20 minutes
  Arms: Study Drug
Drug: Placebo — Prochlorperazine 10 mg administered as an intravenous push over 2 minutes followed by placebo (normal saline)
  Arms: Control Arm

SUMMARY:
The purpose of this research study is to find out if using magnesium in addition to prochlorperazine will help reduce your migraine pain.

DETAILED DESCRIPTION:
The purpose of this prospective, randomized, double-blinded study is to compare the relative efficacy and safety of intravenous magnesium in conjunction with intravenous prochlorperazine in the treatment of migraines. Participants will be patients presenting to the Emergency Department with primary diagnosis of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older
* Able to provide informed consent
* English speaking
* Primary diagnosis of migraine. Patient with a previous diagnosis of migraine, who experience headaches with typical migraine features (e.g at least 2-3 of the following: recurrent, unilateral, pounding or throbbing in nature, associated with nausea), AND with a clinical exclusion of migraine mimics

Exclusion Criteria:

* Pregnancy defined as a positive urine HCG
* Allergy or sensitivity to study drug
* Stated history of renal insufficiency
* Documented history of myasthenia gravis
* Consumption of study drug within 48 hours prior to enrollment
* Previously enrolled in this trial during a different patient encounter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mean change in pain - baseline to 30 minutes | Baseline to 30 minutes after initiation of infusion
  Change in pain score 30 minutes after initiation of infusion. Pain score is measured on a 0-11 point pain intensity numerical rating scale where 0=no pain and 10=worst possible pain.

SECONDARY OUTCOMES:
Mean change in pain - baseline to 45 minutes and baseline to 60 minutes | Baseline to 45 minutes and 60 minutes after initiation of infusion
  Change in pain score 45 minutes and 60 minutes after initiation of infusion. Pain score is measured on a 0-11 point pain intensity numerical rating scale where 0=no pain and 10=worst possible pain.
Number of adverse events | Infusion through hour 2
  Number of adverse events related to study drug within first 2 hours of study drug infusion. Adverse events include hypotension, flushing, akathisia, dystonia, nausea/vomiting, dizziness, drowsiness.
Emergency Department length of stay | Hour 24
  Total time spent in emergency department up until discharge
Number of patients that require rescue medications | Infusion through hour 2
  Number of patients that require administration of rescue meds, which include acetaminophen, NSAIDs, or additional antidopaminergic agents, given within first 2 hours after infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan McKillip, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Christ Medical Center Emergency Department, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No